CLINICAL TRIAL: NCT02108951
Title: A Multicenter, Single Arm Study to Assess Efficacy and Safety of Nilotinib 300mg Twice Daily in Patients With Philadelphia Positive Chronic Myeloid Leukemia in Chronic Phase (Ph+ CML-CP) Who Are Intolerant to Prior Tyrosine Kinase Inhibitors (TKIs).
Brief Title: Study to Assess Efficacy and Safety of Nilotinib 300mg Twice Daily in Patients With Philadelphia Positive Chronic Myeloid Leukaemia (CML) in Chronic Phase Who Are Intolerant to Prior Tyrosine Kinase Inhibitors.
Acronym: ENESTswift
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study was terminated because of slow recruitment
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAMN107AAU04
Record Dates: First submitted 2014-04-07; First posted 2014-04-09 (Estimated); Results first posted 2017-10-27 (Actual); Last update posted 2017-10-27 (Actual); Status verified 2017-09

CONDITIONS: Philidelphia Positive Chronic Myeloid Leukaemia
Keywords: CML; Ph-CML; leukaemia; leukemia; chronic myeloid leukemia; chronic myeloid leukaemia; TKI intolerance; tyrosine kinase inhibitor; tyrosine kinase inhibitor intolerance
MeSH Terms: conditions — Leukemia; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — nilotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Nilotinib (Experimental): Nilotinib was administered orally at 300 mg BD at approximately 12 hour intervals which had to be taken without food. The capsules were to be swallowed whole with water and no food should have been consumed for at least 2 hours before and at least 1 hour after the dose was taken. Prior to the first dose of nilotinib, patients were required to have an imatinib or dasatinib washout period of at least 3 days. Therapy with nilotinib was to be continued for up to 24 months while on study.
  Interventions: Drug: Nilotinib

INTERVENTIONS:
Drug: Nilotinib — Nilotinib 150mg hard gelatin capsules taken orally
  Other Names: AMN107

SUMMARY:
The purpose of this Australian study was to assess the efficacy and safety of nilotinib 300mg twice daily in patients with chronic myeloid leukemia chronic phase who were intolerant but responsive to 1st line treatment with imatinib or dasatinib. Eligible patients have been previously treated with imatinib or dasatinib for at least 3 months and are experiencing non-hematologic toxicity whilst having documented responses that meet PBS authority for 1st line treatment of CML without current MR4.5.

DETAILED DESCRIPTION:
The study was planned to enroll 130 patients to achieve the sample size requirement for a meaning full conclusion. Study got terminated with 20 patients because of slow recruitment. Therefore, due to small sample size, the results cannot be considered clinical significant.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent prior to screening procedures
2. Eastern Cooperative Oncology Grou (ECOG) Performance Status of 0, 1, or 2.
3. Patient with diagnosis of Ph+ CML-CP associated with BCR-ABL quantifiable by RQ-PCR (IS).
4. Patient has received a minimum of 3 months of imatinib or dasatinib treatment (any dose) since initial diagnosis with a documented response.
5. Patient is eligible for Pharmaceutical Benefits Scheme (PBS) reimbursed 1st line TKI treatment.
6. Patient has experienced non-hematological Adverse Events (AE(s)) of any grade, which persisted for at least 1 month despite supportive care or recurred at any grade at least once. Patients who, at the Investigator's discretion, require immediate discontinuation due to the severity of the adverse event are also eligible.
7. No other current or planned anti-leukemia therapies.
8. Adequate organ function.
9. Potassium, Magnesium and Total Calcium above Lower limit of normal.
10. life expectancy of more than 12 months in the absence of any intervention

Key Exclusion Criteria:

1. Prior treatment with nilotinib.
2. Prior Accelerated Phase (AP), Blast Crisis (BC) or allogeneic-transplant (unless the patient received an autologous transplant and was in Chrionic Phase (CP) prior to transplant and never in AP or BC).
3. Patient has documented Molecular Response (MR) 4.5 at the time of study entry
4. Patients with atypical BCR-ABL transcript not quantifiable by standard RQ-PCR.
5. Known impaired cardiac function.
6. Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of study drug.
7. Pregnant or breast feeding (lactating) women.
8. Women of child-bearing potential unwilling or unable to use highly effective contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-07-07 (Actual); Primary Completion 2016-08-10 (Actual); Study Completion 2016-08-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (14):
- Australia (14):
  - Novartis Investigative Site, Canberra, Australian Capital Territory
  - Novartis Investigative Site, Kingswood, New South Wales
  - Novartis Investigative Site, Kogarah, New South Wales
  - Novartis Investigative Site, Liverpool, New South Wales
  - Novartis Investigative Site, St Leonards, New South Wales
  - Novartis Investigative Site, Douglas, Queensland
  - Novartis Investigative Site, Nambour, Queensland
  - Novartis Investigative Site, South Brisbane, Queensland
  - Novartis Investigative Site, Adelaide, South Australia
  - Novartis Investigative Site, Fitzroy, Victoria
  - Novartis Investigative Site, Geelong, Victoria
  - Novartis Investigative Site, Melbourne, Victoria
  - Novartis Investigative Site, Murdoch, Western Australia
  - Novartis Investigative Site, Nedlands, Western Australia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nilotinib
Started | 20 (Indicates patients in enrolled, full analysis and safety set)
Completed | 4
Not Completed | 16
Not completed — Lost to Follow-up | 1
Not completed — Patient's/guardian's decision | 1
Not completed — Study Terminated by Sponsor | 14

BASELINE CHARACTERISTICS:
Arm/Group | Nilotinib
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.9 (15.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 6

OUTCOME MEASURES:

1. Primary Outcome: Deep Molecular Response (MR4.5) Rate: Percentage of Patients Who Have Achieved a 4.5-log Reduction in BCR-ABL Level Within 24 Month
Description: Deep Molecular Response (MR4.5) rate is defined as the percentage of patients who have achieved a 4.5 -log reduction in Breakpoint cluster region - Abelson murine leukemia (BCR-ABL) levels. BCR-ABL levels are measured in patients by real-time quantitative polymerase chain reaction (RQ-PCR) testing of peripheral blood by the 24 months following the commencement of nilotinib therapy.
  MR4.5 corresponds to a BCR-ABL ratio 0.0032% international scale (IS) using RQ-PCR. If a post-baseline value for BCR-ABL is < 0.1 X the baseline value, the patient were classified as achieving a 1 log reduction in BCR-ABL.
Time Frame: Baseline, 96 weeks (24 months)
Population: The full analysis set (FAS) consists of all patients enrolled into the study.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Nilotinib
Number analyzed (Participants) | 20
Percentage of participants | 50 [27.2 to 72.8]

2. Primary Outcome: Molecular Response (MR4.0) Rate: Percentage of Patients Who Have Achieved a 4.0-log Reduction in BCR-ABL Level Within 12 Months and 24 Months
Description: Molecular Response (MR4.0) rate is defined as the percentage of patients who have achieved a 4-log reduction in BCR-ABL levels at 12 months and 24 months following the commencement of nilotinib therapy. Breakpoint cluster region - Abelson murine leukemia (BCR-ABL) levels are measured in patients by real-time quantitative polymerase chain reaction (RQ-PCR) testing of peripheral blood by the 24 months following the commencement of nilotinib therapy.
  MR4.0 corresponds to a BCR-ABL ratio 0.01% international scale (IS) using RQ-PCR. If a post-baseline value for BCR-ABL is < 0.1 X the baseline value, the patients were classified as achieving a 1 log reduction in BCR-ABL.
Time Frame: Baseline, 48 weeks (12 months), 96 weeks (24 months)
Population: The full analysis set (FAS) consists of all patients enrolled into the study. Analysis of MR4.0 was undertaken on the subgroup of the FAS that was not at MR4.0 at baseline.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Nilotinib
Number analyzed (Participants) | 17
Percentage of participants
  Within 12 months | 65 [38.3 to 85.8]
  Within 24 months | 71 [44.0 to 89.7]

3. Primary Outcome: Major Molecular Response (MMR) Rate: Percentage of Patients Who Have Achieved a 3 Log Reduction in BCR-ABL Levels Within 12 Months and 24 Months
Description: Major Molecular Response (MMR) rate is defined as the percentage of patients who have achieved a 3 log reduction in BCR-ABL levels at 12 months and at 24 months following the commencement of nilotinib therapy. Breakpoint cluster region - Abelson murine leukemia (BCR-ABL) levels are measured in patients by real-time quantitative polymerase chain reaction (RQ-PCR) testing of peripheral blood at the 12 and 24 months following the commencement of nilotinib therapy. MMR corresponds to a BCR-ABL ratio 0.1% international scale (IS) using RQ-PCR. If a post-baseline value for BCR-ABL is < 0.1 * the baseline Value, the patient will be classified as achieving a 1 log drop.
Time Frame: Baseline, 48 weeks (12 months), 96 weeks (24 months)
Population: The full analysis set (FAS) consists of all patients enrolled into the study.Analysis of MMR was undertaken on the subgroup of the FAS that was not at MMR at baseline.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Nilotinib
Number analyzed (Participants) | 8
Percentage of participants
  Within 12 months | 75 [34.9 to 96.8]
  Within 24 months | 75 [34.9 to 96.8]

4. Primary Outcome: Duration of Prior TKI Therapy for Patients Based on MR4.5 Achievement Status Within 24 Months
Description: Breakpoint cluster region - Abelson murine leukemia (BCR-ABL) levels are measured in patients by real-time quantitative polymerase chain reaction (RQ-PCR) testing of peripheral blood by the 24 months following the commencement of nilotinib therapy.
  Deep molecular response (MR4.5) rate was defined as the percentage of patients who have achieved a 4.5-log reduction (MR4.5) in BCR-ABL levels during the 24 months following the commencement of nilotinib therapy. MR4.5 corresponds to a BCR-ABL ratio 0.0032% IS using RQ-PCR. If a post-baseline value for BCR-ABL is < 0.1 X the baseline value, the patient were classified as achieving a 1 log reduction in BCR-ABL.
Time Frame: Baseline, 96 weeks (24 months)
Population: The full analysis set (FAS) consists of all patients enrolled into the study.
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Nilotinib
Number analyzed (Participants) | 20
months
  Achieved MR4.5: number analyzed (Participants) | 10
  Achieved MR4.5 | 56.1 (42.06)
  Did not achieve MR4.5: number analyzed (Participants) | 10
  Did not achieve MR4.5 | 45.9 (47.81)

5. Primary Outcome: Number of Patients With MR4.5 Response by Baseline BCR-ABL Response Level Within 24 Months
Description: as for outcome 1
Time Frame: Baseline, 96 weeks (24 months)
Population: The full analysis set (FAS) consists of all patients enrolled into the study. 'n' in categories indicates patients achieved or did not achieve MR4.5 during 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Nilotinib
Number analyzed (Participants) | 20
Participants
  MR4.5 achieved (n=10): No response at baseline: number analyzed (Participants) | 10
  MR4.5 achieved (n=10): No response at baseline | 3
  MR4.5 achieved : MMR at baseline: number analyzed (Participants) | 10
  MR4.5 achieved : MMR at baseline | 4
  MR4.5 achieved : MR4.0 at baseline: number analyzed (Participants) | 10
  MR4.5 achieved : MR4.0 at baseline | 1
  MR4.5 achieved: MR4.5 at baseline: number analyzed (Participants) | 10
  MR4.5 achieved: MR4.5 at baseline | 2
  MR4.5 not achieved: No response at baseline: number analyzed (Participants) | 10
  MR4.5 not achieved: No response at baseline | 5
  MR4.5 not achieved: MMR at baseline: number analyzed (Participants) | 10
  MR4.5 not achieved: MMR at baseline | 5
  MR4.5 not achieved: MR4.0 at baseline: number analyzed (Participants) | 10
  MR4.5 not achieved: MR4.0 at baseline | 0
  MR4.5 not achieved: MR4.5 at baseline: number analyzed (Participants) | 10
  MR4.5 not achieved: MR4.5 at baseline | 0

6. Secondary Outcome: Kinetics of Molecular Response: Percentage of Patients With no Response Based on BCR-ABL Over Time After the Switch to Nilotinib
Description: No response corresponds to a BCR-ABL ratio < 0.1% international scale (IS) using Real-time quantitative polymerase chain reaction (RQ-PCR).
Time Frame: Baseline, week 4, 8, 12, 24, 36, 48, 60, 72, 84, 96
Population: Full analysis set. n = number of patients with evaluable data at the defined time point
Measure: Number; unit: percentage of patients
Arm/Group | Nilotinib
Number analyzed (Participants) | 20
percentage of patients
  Baseline : No Response | 40.0
  Week 4: No response: number analyzed (Participants) | 18
  Week 4: No response | 33.3
  Week 8: No response: number analyzed (Participants) | 19
  Week 8: No response | 26.3
  Week 12: No response | 15.0
  Week 24: No response: number analyzed (Participants) | 16
  Week 24: No response | 18.8
  Week 36: No response: number analyzed (Participants) | 15
  Week 36: No response | 6.7
  Week 48: No response: number analyzed (Participants) | 14
  Week 48: No response | 7.1
  Week 60: No response: number analyzed (Participants) | 8
  Week 60: No response | 0.0
  Week 72: No response: number analyzed (Participants) | 5
  Week 72: No response | 0.0
  Week 84: No response: number analyzed (Participants) | 3
  Week 84: No response | 0.0
  Week 96/End of study: No response: number analyzed (Participants) | 18
  Week 96/End of study: No response | 5.6

7. Secondary Outcome: Kinetics of Molecular Response: Percentage of Patients With MMR Based on BCR-ABL Over Time After the Switch to Nilotinib
Description: MMR corresponds to a BCR-ABL ratio 0.1% international scale (IS) using Real-time quantitative polymerase chain reaction (RQ-PCR).
Time Frame: Baseline, week 4, 8, 12, 24, 36, 48, 60, 72 and 96
Population: Full analysis set. n = number of patients with evaluable data at the defined time point
Measure: Number; unit: percentage of patients
Arm/Group | Nilotinib
Number analyzed (Participants) | 20
percentage of patients
  Baseline : MMR | 45.0
  Week 4: MMR: number analyzed (Participants) | 18
  Week 4: MMR | 55.6
  Week 8: MMR: number analyzed (Participants) | 19
  Week 8: MMR | 36.8
  Week 12: MMR | 40.0
  Week 24: MMR: number analyzed (Participants) | 16
  Week 24: MMR | 31.3
  Week 36: MMR: number analyzed (Participants) | 15
  Week 36: MMR | 26.7
  Week 48: MMR: number analyzed (Participants) | 14
  Week 48: MMR | 28.6
  Week 60: MMR: number analyzed (Participants) | 8
  Week 60: MMR | 12.5
  Week 72: MMR: number analyzed (Participants) | 5
  Week 72: MMR | 0.0
  Week 84: MMR: number analyzed (Participants) | 3
  Week 84: MMR | 0.0
  Week 96/End of study: MMR: number analyzed (Participants) | 18
  Week 96/End of study: MMR | 33.3

8. Secondary Outcome: Kinetics of Molecular Response: Percentage of Patients With MR4.0 Based on BCR-ABL Over Time After the Switch to Nilotinib
Description: MR4.0 corresponds to a BCR-ABL ratio 0.01% international scale (IS) using Real-time quantitative polymerase chain reaction (RQ-PCR).
Time Frame: Baseline, week 4, 8, 12, 24, 36, 48, 60, 72, 84, 96
Population: Full analysis set
Measure: Number; unit: percentage of patients
Arm/Group | Nilotinib
Number analyzed (Participants) | 20
percentage of patients
  Baseline : MR4.0 | 5.0
  Week 4: MR4.0: number analyzed (Participants) | 18
  Week 4: MR4.0 | 5.6
  Week 8: MR4.0: number analyzed (Participants) | 19
  Week 8: MR4.0 | 15.8
  Week 12: MR4.0 | 10.0
  Week 24: MR4.0: number analyzed (Participants) | 16
  Week 24: MR4.0 | 18.8
  Week 36: MR4.0: number analyzed (Participants) | 15
  Week 36: MR4.0 | 20.0
  Week 48: MR4.0: number analyzed (Participants) | 14
  Week 48: MR4.0 | 14.3
  Week 60: MR4.0: number analyzed (Participants) | 8
  Week 60: MR4.0 | 12.5
  Week 72: MR4.0: number analyzed (Participants) | 5
  Week 72: MR4.0 | 60.0
  Week 84: MR4.0: number analyzed (Participants) | 3
  Week 84: MR4.0 | 33.3
  Week 96/End of study: MR4.0: number analyzed (Participants) | 18
  Week 96/End of study: MR4.0 | 16.7

9. Secondary Outcome: Kinetics of Molecular Response: Percentage of Patients With MR4.5 Based on BCR-ABL Over Time After the Switch to Nilotinib
Description: MR4.5 corresponds to a BCR-ABL ratio 0.0032% international scale (IS) using Real-time quantitative polymerase chain reaction (RQ-PCR).
Time Frame: Baseline, week 4, 8, 12, 24, 36, 48, 60, 72, 84, 96
Population: Full analysis set. n = number of patients with evaluable data at the defined time point
Measure: Number; unit: percentage of patients
Arm/Group | Nilotinib
Number analyzed (Participants) | 20
percentage of patients
  Baseline : MR4.5 | 10.0
  Week 4: MR4.5: number analyzed (Participants) | 18
  Week 4: MR4.5 | 5.6
  Week 8: MR4.5: number analyzed (Participants) | 19
  Week 8: MR4.5 | 21.1
  Week 12: MR4.5 | 35.0
  Week 24: MR4.5: number analyzed (Participants) | 16
  Week 24: MR4.5 | 31.3
  Week 36: MR4.5: number analyzed (Participants) | 15
  Week 36: MR4.5 | 46.7
  Week 48: MR4.5 | 50.0
  Week 60: MR4.5: number analyzed (Participants) | 8
  Week 60: MR4.5 | 75.0
  Week 72: MR4.5: number analyzed (Participants) | 5
  Week 72: MR4.5 | 40.0
  Week 84: MR4.5: number analyzed (Participants) | 3
  Week 84: MR4.5 | 66.7
  Week 96/End of study: MR4.5: number analyzed (Participants) | 18
  Week 96/End of study: MR4.5 | 44.4

10. Secondary Outcome: Kaplan-Meier Estimates of Time to Deep Molecular Response (MR4.5)
Description: Breakpoint cluster region - Abelson murine leukemia (BCR-ABL) levels is measured in patients by real-time quantitative polymerase chain reaction (RQ-PCR) testing of peripheral blood by the 24 months following the commencement of nilotinib therapy. MR4.5 corresponds to a
  BCR-ABL ratio 0.0032% IS using RQ-PCR. The derivation of time to molecular response for patients in the study was measured from the date of first nilotinib use, defined as follows:
  Days to MR4.5 = date of assessment where BCR-ABL ratio is 0.0032% IS - date of baseline + 1.
Time Frame: 96 weeks (24 months)
Population: The full analysis set (FAS) consists of all patients enrolled into the study. N represents all patients in FAS who achieved MR4.5.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Nilotinib
Number analyzed (Participants) | 10
days | 343 [64 to NA] — Upper limit is not estimable due to the low number of patients achieving MR4.5.

11. Secondary Outcome: Time to Progression-free Survival (PFS)
Description: PFS was defined as the time from the date of baseline visit to the date of earliest progression-defining event: namely progression (or withdrawal due to progression to blast crisis (BC) or accelerated phase (AP) disease), or death from any cause.
  Patients who did not progress were censored at earliest of the following:
  * the date of the 24-month visit;
  * the date of loss to follow-up;
  * the date of discontinuation of study treatment for any reason other than progression to BC, or AP disease, or death
Time Frame: 96 weeks (24 months)
Population: The FAS consists of all patients enrolled into the study. There were no withdrawals due to progression to BC or AP disease, and there were no recorded deaths during the study.
Arm/Group | Nilotinib
Number analyzed (Participants) | 0

12. Secondary Outcome: Time to Event Free Survival (EFS)
Description: EFS was defined as the time from date of baseline visit to the first occurrence of any of the following: Disease progression, treatment failure or death from any cause, whichever was earlier. Patients who did not have an event of interest were censored at earliest of the following:
  * the date of the 24-month visit;
  * the date of loss to follow-up;
  * the date of withdrawal from the study for any reason other than lack of efficacy/progressive disease, tolerance to reduced dose or death
Time Frame: 96 weeks (24 months)
Population: There were no patients in the study who were recorded as experiencing treatment failure.
Arm/Group | Nilotinib
Number analyzed (Participants) | 0

13. Secondary Outcome: Number of Patients With Events Reported at Baseline That Have Shown an Improvement in Non-hematological AE Severity Compared to Week 12 Visit
Description: The total number of patients that have showed improvement with respect to CTCAE grades at the time of the 12-week visit are reported. Improved is defined as prior to, or at the time of the 12-week visit, the AE has completely resolved.
Time Frame: Baseline, week 12 (month 3)
Population: The Safety Set (SS) consisted of all patients in the FAS who received at least 1 dose of study drug and had at least 1 post-baseline safety assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Nilotinib
Number analyzed (Participants) | 20
Participants
  Improved : Yes | 11
  Improved: No | 9

14. Secondary Outcome: Mean M.D. Anderson Symptom Inventory - Chronic Myeloid Leukemia (MDASI-CML)
Description: Quality of life was assessed using the M.D. Anderson Symptom Inventory - Chronic Myeloid Leukemia (MDASI-CML) self-administered questionnaire for adult CML patients. The questionnaire consisted of 13 core questions in part I measuring the severity of symptoms, 6 questions in part 2 assessing the interference of symptoms on daily living. The CML component of the MDASI provided an additional 7 CML-specific symptom items: diarrhea, swelling, rash/skin change, muscle soreness/cramping, bruising/bleeding easily, malaise, and headache. In part I (13 questions) and the CML component (7 questions) each question was scored from 0 to 10 where 0 indicates a symptom is not present and 10 indicate the symptom is "as bad as you can imagine". For part 1 the total score can therefore range from 0 to 130 and for CML 0 to 70. Part 2 is also recorded on a 0 to 10 scale, but 0 now indicates that the symptom "did not interfere" and 10 "interfered completely". The total score can range from 0 to 60.
Time Frame: Baseline, week 12, 24, 48, 96
Population: The full analysis set (FAS) consists of all patients enrolled into the study. 'n' in the categories represents the number of patients with evaluable data for MDASI part 1/MDASI part 2/CML component at different time points. Week 96 includes end of study results for patients that did not complete the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Nilotinib
Number analyzed (Participants) | 20
units on a scale
  Baseline: MDASI part 1 | 26.6 (23.88)
  Week 12: MDASI part 1: number analyzed (Participants) | 19
  Week 12: MDASI part 1 | 22.7 (20.31)
  Week 24: MDASI part 1: number analyzed (Participants) | 16
  Week 24: MDASI part 1 | 20.7 (18.08)
  Week 48: MDASI part 1: number analyzed (Participants) | 12
  Week 48: MDASI part 1 | 20.4 (16.57)
  Week 96: MDASI part 1: number analyzed (Participants) | 19
  Week 96: MDASI part 1 | 17.5 (20.44)
  Baseline: MDASI part 2 | 12.4 (14.17)
  Week 12: MDASI part 2: number analyzed (Participants) | 18
  Week 12: MDASI part 2 | 7.8 (11.92)
  Week 24: MDASI part 2: number analyzed (Participants) | 16
  Week 24: MDASI part 2 | 8.2 (12.20)
  Week 48: MDASI part 2: number analyzed (Participants) | 12
  Week 48: MDASI part 2 | 7.6 (10.53)
  Week 96: MDASI part 2 | 9.9 (15.59)
  Baseline: CMLcomponent | 40.9 (35.02)
  Week 12: CMLcomponent: number analyzed (Participants) | 18
  Week 12: CMLcomponent | 31.5 (30.10)
  Week 24: CMLcomponent: number analyzed (Participants) | 16
  Week 24: CMLcomponent | 30.8 (28.62)
  Week 48: CMLcomponent: number analyzed (Participants) | 12
  Week 48: CMLcomponent | 28.2 (24.43)
  Week 96 CMLcomponent: number analyzed (Participants) | 19
  Week 96 CMLcomponent | 25.4 (31.06)

ADVERSE EVENTS:
Time Frame: Adverse Events are collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV). All Adverse events are reported in this record from First Patient First Treatment until Last Patient Last Visit.
Arm/Group | Nilotinib
Serious Adverse Events (participants affected / at risk) | 1/20
Other Adverse Events (participants affected / at risk) | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nilotinib (N=20)
Pneumonia (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nilotinib (N=20)
Constipation (Gastrointestinal disorders) | 4
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4
Fatigue (General disorders) | 11
Influenza like illness (General disorders) | 2
Lower respiratory tract infection (Infections and infestations) | 2
Nasopharyngitis (Infections and infestations) | 2
Upper respiratory tract infection (Infections and infestations) | 4
Urinary tract infection (Infections and infestations) | 3
Alanine aminotransferase increased (Investigations) | 2
Blood alkaline phosphatase increased (Investigations) | 2
Blood bilirubin increased (Investigations) | 2
Gamma-glutamyltransferase increased (Investigations) | 4
Weight decreased (Investigations) | 2
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Eczema (Skin and subcutaneous tissue disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 3

LIMITATIONS AND CAVEATS:
The study was planned to enroll 130 patients. Study got terminated with 20 patients because of slow recruitment. Therefore, due to small sample size, the results cannot be considered clinical significant.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.